CLINICAL TRIAL: NCT02322242
Title: Comparison of the Effects of Perineural Versus Systemic Dexamethasone on Low Dose Interscalene Brachial Plexus Block: A Randomized Control Trial
Brief Title: The Effects of Dexamethasone on Low Dose Interscalene Brachial Plexus Block
Acronym: ISB-Dex
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dr. Stephen Choi (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Sponsor-Investigator, Dr. Stephen Choi, Assistant Professor and Staff Anesthetist, Department of Anesthesia, Sunnybrook Health Sciences Centre
Organization: Sunnybrook Health Sciences Centre (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 437-2013
Record Dates: First submitted 2014-12-16; First posted 2014-12-23 (Estimated); Results first posted 2020-07-07 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Shoulder Surgery; Nerve Block
MeSH Terms: interventions — dexamethasone 21-phosphate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Perineural Dexamethasone (Active Comparator): ISB performed with local anesthetic (ropivacaine 0.5%) and perinerual dexamethasone (4mg)
  Interventions: Drug: Perineural dexamethasone
- Systemic Dexamethasone (Other): ISB with local anesthetic alone (ropivacaine 0.5%) alone and intravenous dexamethasone (4mg)
  Interventions: Drug: Systemic Dexamethasone

INTERVENTIONS:
Drug: Systemic Dexamethasone — Intravenous infusion of dexamethasone (4mg)
  Other Names: Dexamethasone Sodium Phosphate Injection
  Arms: Systemic Dexamethasone
Drug: Perineural dexamethasone — Perinerual administration of dexamethasone (4mg)
  Other Names: Dexamethasone Sodium Phosphate Injection
  Arms: Perineural Dexamethasone

SUMMARY:
A standard interscalene nerve block is performed with long acting local anesthetic (bupivacaine or ropivacaine in concentrations varying from 0.25% to 0.75%). The purpose of this study is to investigate the effect of the addition of perineural dexamethasone (4mg) to a standard ropivacaine solution (0.5%) on analgesic duration of low dose interscalene block compared to ropivacaine alone for interscalene block with systemic dexamethasone.

Ropivacaine is not an intervention as a local anesthetic is pre-requisite to performing a nerve block.

DETAILED DESCRIPTION:
Interscalene brachial plexus block (ISB) is regarded as the standard of care for analgesia after shoulder surgery providing superior analgesia and reducing opioid consumption. Shoulder surgery, previously requiring inpatient admission for pain control, is now commonly performed on an ambulatory basis facilitated by ISB analgesia. The effects of single injection ISB dissipate after several hours unmasking the moderate to severe pain of the surgical insult and require strong opioid analgesia. Efforts to prolong ISB duration by increasing local anaesthetic (LA) dose are limited by their pharmacodynamics and narrow therapeutic window. To address some of these issues faced with prolonging ISB analgesia the addition of perineural adjuvants to local anesthetic (eg. clonidine, dexmedetomidine), have been investigated in an attempt to prolong peripheral nerve block duration with limited success. However, the corticosteroid dexamethasone, has been added to local anesthetic solutions for ISB and has demonstrated promise in preliminary studies. Perineural dexamethasone (8-10mg) in conjunction with local anesthetic prolongs the duration of ISB with an effect sizes ranging from 40% to 75% (absolute effect ~ 6 to 10 hours). Dexamethasone, however, is only approved for intramuscular or intravenous administration and therefore perineural use is currently off-label. There are several reasons that warrant a new randomized trial. Chiefly, all of the previous trials do not reflect modern regional anesthetic practice. These trials utilized peripheral nerve stimulation (PNS) and local anesthetic volumes of 30 to 40 ml. Modern ultrasound guided ISB (US-ISB) allows for more accurate, targeted deposition of local anesthetic with volumes ranging from 5 to 10 ml with no difference in block efficacy or duration compared to larger volumes (≥20ml). An ideal solution would be a local anesthetic with adjuvant mixture that allowed administration of lower volumes but with prolonged analgesic duration. The use of low dose local anesthetic with dexamethasone could be one such solution. A trial that demonstrates enhanced block quality and duration associated with perineural dexamethasone added to low dose local anesthetic may allow us to achieve both prolonged duration of effect and reduced side effects due to unwanted local anesthetic spread. This would create further significant benefits for patients and further promote the use of low dose local anesthetic techniques to anesthesiologists who do not currently use this technique.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing arthroscopic shoulder surgery at Sunnybrook Health Sciences Centre, Toronto Western Hospital and Women's College Hospital.
2. ASA functional status class I to III
3. Age 18 to 80 years
4. BMI ≤ 35 kg/m2

Exclusion Criteria:

1. Lack of patient consent
2. Allergy to dexamethasone or ropivacaine
3. BMI > 35 kg/m2
4. Contraindications to low dose dexamethasone including peptic ulcer disease, systemic infection, glaucoma, active varicella/herpetic infections, diabetes mellitus
5. Contraindications to ISB including severe Chronic Obstructive Pulmonary Disease (Forced expiratory volume < 40% predicted), coagulopathy, pre-existing neurologic deficit in ipsilateral upper extremity, localized infection
6. Pregnant or nursing females
7. Chronic opioid use defined as > 30mg oral morphine or equivalent per day
8. Unable to take acetaminophen or celecoxib

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Choi, MD,FRCPC,MSc, Principal Investigator — SunnybrookHealth Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McHardy PG, Singer O, Awad IT, Safa B, Henry PDG, Kiss A, Au SK, Kaustov L, Choi S. Comparison of the effects of perineural or intravenous dexamethasone on low volume interscalene brachial plexus block: a randomised equivalence trial. Br J Anaesth. 2020 Jan;124(1):84-91. doi: 10.1016/j.bja.2019.08.025. Epub 2019 Oct 5. PMID 31591018

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment setting: pre-operative anesthesia clinic 182 recruited because of time lag between recruitment and surgery
Period: Overall Study
Arm/Group | Perineural Dexamethasone | Systemic Dexamethasone
Started | 92 | 90
Primary Outcome | 92 | 90
1 Week Follow-up | 90 (2 lost to follow-up for secondary outcomes) | 89 (1 lost to follow-up for secondary outcomes)
Completed | 92 | 90
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Perineural Dexamethasone | Systemic Dexamethasone | Total
Number analyzed (Participants) | 92 | 90 | 182
Age, Continuous [Mean (Full Range); unit: years] | 51.6 [18 to 73] | 52.8 [22 to 76] | 52.2 [18 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 21 | 46
  Male | 67 | 69 | 136
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Duration of Sensory Block
Description: Defined as time from completion of block procedure to NRS for pain > 0 (in hours)
Time Frame: 1 day postoperative
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Perineural Dexamethasone | Systemic Dexamethasone
Number analyzed (Participants) | 92 | 90
minutes | 521 (442) | 566 (428)

2. Secondary Outcome: Time to First Opioid Consumption
Description: Defined as time from completion of block procedure to first consumption of opioid analgesic (in hours)
Time Frame: 1 day postoperative
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Perineural Dexamethasone | Systemic Dexamethasone
Number analyzed (Participants) | 92 | 90
hours | 9.1 (6.9) | 9.6 (10.8)

3. Secondary Outcome: Duration of Motor Block
Description: Defined as time from completion of block procedure to return to baseline motor function (in hours)
Time Frame: 1 day postoperative
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Perineural Dexamethasone | Systemic Dexamethasone
Number analyzed (Participants) | 92 | 90
hours | 18.5 (13.8) | 20.3 (22.3)

4. Secondary Outcome: Post-operative Oxygen Saturation on Room Air
Description: Pulse oximetry (in %) measured 1 hour after arrival in post-operative recovery room, scale 0-100, higher number is better
Time Frame: 1 hour postoperative
Measure: Mean (Standard Deviation); unit: Room air oxygen saturation percent
Arm/Group | Perineural Dexamethasone | Systemic Dexamethasone
Number analyzed (Participants) | 92 | 90
Room air oxygen saturation percent | 96.6 (2.3) | 97.0 (2.4)

5. Secondary Outcome: Opioid Consumption
Description: Opioid consumption (in oral morphine equivalents) will be recorded at 12 hours, 24 hours, and 7 days
Time Frame: 7 days postoperative
Measure: Mean (Standard Deviation); unit: mg (oral morphine equivalent)
Arm/Group | Perineural Dexamethasone | Systemic Dexamethasone
Number analyzed (Participants) | 92 | 90
mg (oral morphine equivalent) | 148.8 (117.9) | 167.2 (140.0)

6. Secondary Outcome: Numeric Rating Scale for Pain (NRS 0-10)
Description: Recorded at 12 hours, 24 hours, and 7 days 0 is no pain, 10 is the worst pain imaginable. Lower number is better.
Time Frame: 7 days postoperative
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Perineural Dexamethasone | Systemic Dexamethasone
Number analyzed (Participants) | 92 | 90
units on a scale
  7 days | 3.1 (2.3) | 3.4 (2.4)
  24hours | 4.9 (2.6) | 4.7 (2.6)
  12hours | 3.3 (3.0) | 3.3 (2.9)

7. Secondary Outcome: Postoperative Serum Blood Glucose
Description: Measured 1 hour after arrival to the post-operative recovery room
Time Frame: 1 hour postoperative
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Perineural Dexamethasone | Systemic Dexamethasone
Number analyzed (Participants) | 92 | 90
mmol/L | 6.8 (1.0) | 6.6 (1.1)

8. Secondary Outcome: Number of Participants With Nerve Damage From Interscalene Block
Description: Defined as persistent paresthesia, and sensory/motor block at 7 days
Time Frame: 7 Days postoperative
Measure: Count of Participants; unit: Participants
Arm/Group | Perineural Dexamethasone | Systemic Dexamethasone
Number analyzed (Participants) | 92 | 90
Participants | 0 | 0

9. Secondary Outcome: Infection
Description: Number of participants with localized infection at nerve block site
Time Frame: 7 Days postoperative
Measure: Count of Participants; unit: Participants
Arm/Group | Perineural Dexamethasone | Systemic Dexamethasone
Number analyzed (Participants) | 92 | 90
Participants | 0 | 0

10. Secondary Outcome: Number of Participants With Postoperative Nausea and/or Vomiting
Description: Number of participants with postoperative nausea and/or vomiting assessed at 12 hours, 24, hours, and 7 days postoperatively
Time Frame: 7 days postoperative
Measure: Count of Participants; unit: Participants
Arm/Group | Perineural Dexamethasone | Systemic Dexamethasone
Number analyzed (Participants) | 92 | 90
Participants | 32 | 32

ADVERSE EVENTS:
Time Frame: Adverse events were recorded over a 1 week follow-up period
Arm/Group | Perineural Dexamethasone | Systemic Dexamethasone
All-Cause Mortality (participants affected / at risk) | 0/92 | 0/90
Serious Adverse Events (participants affected / at risk) | 0/92 | 0/90
Other Adverse Events (participants affected / at risk) | 0/92 | 0/90

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-10-25): https://cdn.clinicaltrials.gov/large-docs/42/NCT02322242/Prot_SAP_000.pdf